CLINICAL TRIAL: NCT02254889
Title: Pain After Endoscopic Submucosal Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gangnam Severance Hospital (Other)
Responsible Party: Principal Investigator, Da Hyun Jung, Doctor, Gangnam Severance Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3-2011-0007
Record Dates: First submitted 2014-09-25; First posted 2014-10-02 (Estimated); Last update posted 2016-02-12 (Estimated); Status verified 2016-02

CONDITIONS: Gastric Neoplasm
MeSH Terms: conditions — Stomach Neoplasms | interventions — Proton Pump Inhibitors

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pre-ESD group (Active Comparator): All subjects were randomly assigned to treatment with intravenous proton pump inhibitor (PPI) before ESD.
  Interventions: Drug: proton pump inhibitor
- post-ESD group (Placebo Comparator): All subjects were randomly assigned to treatment with intravenous proton pump inhibitor (PPI) after ESD.
  Interventions: Drug: proton pump inhibitor

INTERVENTIONS:
Drug: proton pump inhibitor — ). In the pre-ESD therapeutic group, a standard intravenous dose of PPI was given 2 hours before ESD. In the post-ESD therapeutic group, patients also received intravenous PPI in standard doses, once in the evening after ESD.

SUMMARY:
Endoscopic submucosal dissection (ESD) is widely used for local treatment of gastric neoplasms. Although ESD-related complications such as bleeding and perforation have been reported, data is currently lacking on the development of pain, which is one of the most common adverse events after ESD. Therefore, in the present study, we investigated the incidence and clinicopathologic risk factors of pain after ESD.

DETAILED DESCRIPTION:
A prospective randomized controlled study was conducted evaluating 156 patients with gastric neoplasms treated by ESD at Gangnam Severance Hospital between April 2011 and December 2014. All subjects were randomly assigned to treatment with intravenous proton pump inhibitor (PPI) either before or after ESD.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing ESD for gastric neoplasms

Exclusion Criteria:

* (1) history of acid suppressive medication within 1 week prior to the procedure; (2) known gastrointestinal disorders, such as peptic ulcer disease, which might impact epigastric pain assessment; (3) current or regular use of pain medication; (4) history of upper gastrointestinal surgery; (5) multiple lesions requiring ESD; (6) perforation during ESD; and (7) significant cardiovascular, renal, hepatic, neurotic, or psychological disorders

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2011-04; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
A 10-cm VAS was used to evaluate pain after ESD. | Pain was rated at 24 hours after ESD.

CONTACTS AND LOCATIONS:
Overall Officials: Young Hoon Youn, MD, PhD, Study Director — Gangnam Severance Hospital
Locations (1):
- Da Hyun Jung, Seoul, South Korea

REFERENCES:
- [Derived] Jung DH, Youn YH, Kim JH, Park H. Factors influencing development of pain after gastric endoscopic submucosal dissection: a randomized controlled trial. Endoscopy. 2015 Dec;47(12):1119-23. doi: 10.1055/s-0034-1392537. Epub 2015 Jul 10. PMID 26165736